CLINICAL TRIAL: NCT05887687
Title: A Study to Evaluate 68Ga-P3 PET/CT Imaging of PSMA Expression in Malignant Tumors
Brief Title: 68Ga-P3 PET/CT Imaging in Malignancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xing YANG, Principal Investigator, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: [68Ga]P3
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Neoplasms
Keywords: [68Ga]P3; PSMA; PET/CT; Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]P3 (Experimental): Subjects with suspected or confirmed malignancy will receive an intravenous injection of 68Ga-P3 followed by PET imaging. The subjects will also receive a whole-body 18F-FDG PET/CT scan within a one-week period.
  Interventions: Drug: [68Ga]P3

INTERVENTIONS:
Drug: [68Ga]P3 — 68Ga-P3 is injected intravenously with a dose of 0.06-0.08 mCi/kg.
  Other Names: [68Ga]-P3; PSMA specific PET imaging

SUMMARY:
Prostate-specific membrane antigen (PSMA) is a type II transmembrane glycoprotein that consists of 750 amino acids. It is highly expressed on most prostate cancer cells and neovascular endothelial cells of tumors, making PSMA a highly specific and significant imaging target for malignancies.

[68Ga]P3, a novel molecular probe of PET imaging agent that targets PSMA, can be used in the diagnosis and research of a wide variety of PSMA high-expression malignanciesr.

DETAILED DESCRIPTION:
Prostate-specific membrane antigen (PSMA) is a type II transmembrane glycoprotein that consists of 750 amino acids. It is highly expressed on most prostate cancer cells and neovascular endothelial cells of tumors, making PSMA a highly specific and significant imaging target for malignancies.[68Ga]P3, a novel molecular probe of PET imaging agent that targets PSMA, can be used in the diagnosis and research of a wide variety of PSMA high-expression malignanciesr.

ELIGIBILITY:
Inclusion Criteria:

patients with confirmed or suspected cancer; 18F-FDG PET/CT within 1 week; Signed written informed consent

Exclusion Criteria:

Pregnant and lactating women; Female patients plan to become pregnant within 6 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficacy of 68Ga-P3 PET/CT in the evaluation of malignant tumors | 1 year
  Compare the standardized Uptake Value (SUV) of lesions on 68Ga-P3 and 18F-FDG PET/CT
The detection efficacy of 68Ga-P3 PET/CT in the evaluation of malignant tumors | 1 year
  Compare the number of lesions detected by 68Ga-P3 and 18F-FDG PET/CT, based on the pathology or clinical follow-up as gold standard.

SECONDARY OUTCOMES:
The dosimetry of 68Ga-P3 | 1 year
  Research on the dose distribution of 68Ga-P3 in healthy volunteers and cancer patients by 1-hour dynamic PET/CT acquisition and analyze by the dosimetry software
Quantitative evaluation of 68Ga-P3 | 1 year
  Evaluation of quantitative parameters of 68Ga-P3, such as time-activity curve.
Correlation with pathological expression | 1 year
  Analyze PSMA expression at the imaging level in combination with PSMA expression in pathological specimens

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China